CLINICAL TRIAL: NCT06714110
Title: A Retrospective Review of Clinical and Radiographic Outcomes Following the Use of the Precice Intramedullary Limb Lengthening (IMLL) System in Pediatric Limb Lengthening Procedures
Brief Title: A Review of Precice Intramedullary Limb Lengthening (IMLL) System for Limb Lengthening Procedures in Children.
Status: Enrolling by invitation | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.ILL0723
Record Dates: First submitted 2024-11-07; First posted 2024-12-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Limb Length Discrepancy
Keywords: Precice IMLL; external fixator; Limb length discrepancy surgery; index bone; femur; tibia; surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Precice IMLL System: Patients 12 years of age or younger received Precice IMLL for correction of limb length discrepancy.
  Interventions: Device: Intramedullary Limb Lengthening Device
- External Fixator: Patients 12 years of age or younger received an external fixator for correction of limb length discrepancy.
  Interventions: Device: External Fixator Limb Lengthening Device

INTERVENTIONS:
Device: Intramedullary Limb Lengthening Device — The Precice IMLL System is composed of the Precice nail, screws, and uses an external remote controller (ERC) for rod distraction. The Precice IMLL System is designed to fit the anatomy of long bones and is intended to be placed internally in an intramedullary manner. It achieves limb correction through gradual lengthening or compression and providing intramedullary fixation for fractures of long bones.
  Groups: Precice IMLL System
Device: External Fixator Limb Lengthening Device — External fixator devices consist of an external frame (ring, half-ring, monolateral, and rail); bone fixation is accomplished by the transcutaneous bone fixations implants (pins, wires, cables, screws), and the lengthening is accomplished by the vertical components (struts). Generally, femoral lengthening devices are monolateral and tibial lengthening devices have ring or half-ring frames. The external fixators are made of a variety of materials, including stainless steel, titanium, carbon fiber, and aluminum.
  Groups: External Fixator

SUMMARY:
This study will look at how safe and effective limb lengthening surgeries are for the femur and tibia in children 12 years old and younger. We will examine any complications from the surgery, the results of X-rays, and feedback from patients. The study will involve the Precice Intramedullary Limb Lengthening (IMLL) System and external fixator devices for limb lengthening.

DETAILED DESCRIPTION:
As a retrospective chart review, all patients involved in this study will have undergone surgery for their limb length discrepancy according to the standard of care of the practitioner using either the Precice IMLL or an external fixator. Under this protocol, available patient outcomes, plain radiographs, and complications will be obtained from the existing medical records of all eligible index surgeries. An index surgery is defined as the first limb lengthening surgery performed by a study investigator on the index bone with either the Precice IMLL or an external fixator. Each patient may have up to 4 eligible index surgeries (right and left femur, right and left tibia) and be included in both the Precice IMLL and external fixator groups.

ELIGIBILITY:
Inclusion Criteria:

* All potential index surgeries must meet the inclusion criteria below in order to be considered for enrollment:

  1. Patient was 12 years of age or younger at the time of the index surgery.
  2. Diagnosis of femoral or tibial limb length discrepancy greater than or equal to 2.0 cm.
  3. Limb length discrepancy secondary to congenital or acquired etiologies.
  4. Patients received limb lengthening treatment of the femur or tibia with the Precice IMLL System or an external fixator limb lengthening device.
  5. Minimum medullary canal diameter ≥6 mm in the treated bone - Precice IMLL System treatment group only.
  6. Closed or nonfunctioning physeal growth plates in the treated bone - Precice IMLL System treatment group only.
  7. Minimum of 12 months of follow-up.
  8. Available medical and radiographic records preoperatively through consolidation.

Exclusion Criteria:

* Index surgeries will be excluded from consideration for the study if they meet any of the following criteria:

  1. Patients with unresolved limb lengthening-related adjacent joint contractures (loss of range of motion), subluxation, or dislocation prior to the index surgical procedure.
  2. Patients with uncorrected coronal or sagittal plane angular malalignment following the index surgical procedure.
  3. Patients with unresolved complications related to previous limb lengthening on the index or different limbs, including unhealed pin sites and/or residual bone infection (from external fixator devices) on the index limb.
  4. Patients with femoral head osteonecrosis from a previous implantation of a femoral nail prior to the index surgical procedure.
  5. Patients with a previous implantation of a femoral or tibial nail across an open physeal growth plate prior to the index surgical procedure.

Ages: 0 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric (12 years and under) population
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Bone (femur or tibia) lengthening | At least 1 yr post-op
  Achievement of targeted limb length
Osteotomy Healing | At least 1 yr post-op
  Assessment of osteotomy healing using the following descriptors:
  * Premature healing: Defined as osteotomy healing before the target length is achieved.
  * Healed (consolidated): Defined as the presence of full corticalization (ossified) of regenerate bone of three of four cortices seen on AP and lateral radiographs.
  * Delayed union (consolidation): Defined as bone union taking greater than 6 months but with progressive improvement on radiographs and the osteotomy eventually healed.
  * Partial union (consolidation): Defined as incomplete bone healing, i.e., radiographic healing at only 1 or 2 cortices on AP and lateral views.
  * Nonunion (pseudarthrosis): Defined as lack of complete healing within 6 months of the end of the lengthening period.
Frequency of device related complications | Post-op through at least 1 year post-op
  Review of investigator-reported device-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, Study Director — Globus Medical
Locations (1):
- Paley Institute, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No